CLINICAL TRIAL: NCT01732679
Title: A Prospective Multicenter Study of Stroke Rehabilitation in Seven Countries: Norway, China, USA, Russia, Israel, Palestine, and Sweden.
Brief Title: Sunnaas International Network´s Stroke Study
Acronym: SINs
Status: Completed | Type: Observational
Sponsor: Sunnaas Rehabilitation Hospital (Other)
Collaborators: China Rehabilitation Research Center (Other Government); Sichuan 81 Rehabilitation Center, Chengdu (Unknown); NYU Langoon medical center; The Rusk Institute of Rehabilitation Medicine, New York (Unknown); City outpatient clinics №2,Petrozavodsk, Petrozavodsk (Other); Sheba Medical Center (Other Government); Al-Wafa Rehabilitation Hospital (Other); Bethlehem Arab Society for Rehabilitation, Betlehem (Unknown); Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Birgitta Langhammer, Associate professor/ project manager, Sunnaas Rehabilitation Hospital
Other Study IDs: SINs stroke study
Record Dates: First submitted 2012-11-08; First posted 2012-11-26 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Cerebral Stroke
Keywords: stroke, rehabilitation, multidisciplinary, description
MeSH Terms: conditions — Stroke | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- stroke patients: specialized rehabilitation in a multidisciplinary team, Sunnaas International Network
  Interventions: Other: rehabilitation

INTERVENTIONS:
Other: rehabilitation — Description of specialized rehabilitation and Influence on activities, life satisfaction, psycho social aspects 6 and 12 months post discharge
  Other Names: multidisciplinary specialised rehabilitation

SUMMARY:
A descriptive study of the stroke rehabilitation content in specialized clinics in seven countries: procedures for admission to rehabilitation, services available and provided to patients, as well as duration of the stay and discharge routines. An observational study of changes in regard to the physical function, quality of life and psycho-social factors in stroke patients before and after specialized rehabilitation

DETAILED DESCRIPTION:
The descriptive study is two folded:

1) Description of the rehabilitation centers and the content the respective clinic presents as specialized rehabilitation.

A description of the expected change this input will result in in form of patients change in ADL and life satisfaction, with repeated measurements:

2a) reports of change in activities of daily living from baseline, to one fixed time (18-22 days in rehab),at discharge (which will vary),6 and 12 months post discharge (relatively fixed time) .

2b) reports of possible change in life satisfaction at baseline, discharge, 6 and 12 months after discharge.

Since the times for admission is expected to vary, which will be described under 1),we also want to measure if and how this difference might influence results. Therefore a fixed measure is inserted between admission and discharge. we have added a "relatively" fixed date at 6 months post stroke in order to see if change of function from specialized rehabilitation will differ in a longitudinal perspective, and if possible to see if the difference in time to admission (time from debut till admission in specialized rehabilitation)might influence results.

3) description of psycho- social factors at 6 and 12 months post discharge

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis of stroke, in need of specialized comprehensive rehabilitation, voluntary participation

Exclusion Criteria:

* sub-arachnoid hæmorrhage, tumor or other severe medical condition in combination with stroke that will influence outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stroke patients in need of specialised comprehensive rehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
activities of daily living | patients will be followed 6 months from baseline testing
  Changes in Activities of daily living are monitored as an indirect evaluation of how the specialized rehabilitation may influence patients' outcomes.

SECONDARY OUTCOMES:
The Life Satisfaction checklist (LiSat-11) | patients will be followed 6 months from baseline testing
  LiSat-11 consists of patients estimations of satisfaction with life as a whole as well as satisfaction in ten specific domains: vocation, economy, leisure, contacts, sexual life, activities of daily living (ADL), family life, partner relationship, somatic health, psychological health

OTHER OUTCOMES:
National Institutes of health stroke scale (NIHSS) | patients will be tested baseline and at discharge
  NIHSS is a clinical stroke assessment tool to evaluate and document neurological status in acute stroke patients.
  The timeframe for discharge will vary with the different clinics since this is one of the differences expected.
  Length of stay is one of the outcomes
Modified Rankin Scale | patients will be followed 6 months from baseline testing
  it is an evaluation of the degree of disability or dependence in the daily activities of people who have suffered a stroke
Description of the psycho- social situation | 6 months after discharge
  A semi - structured interview, with focus on the psycho-social situation 6 months after rehabilitation, will be performed. Questions will focus on the work-, financial situation, what sort of follow-up services, recreational- and social activities are available, and what is considered the major change of life after stroke.
description of institution | baseline
  a questionaire where the participants are required to describe the services available, methods used in rehabilitation, intensity of training, procedures for intake and discharge
registration data | baseline
  questionnaire regarding demographic data; age, gender, civil status, comorbidity, medication

CONTACTS AND LOCATIONS:
Overall Officials: Johan K Stanghelle, PhD, MD, Study Director — Sunnaas rehabilitation hospital, University of Oslo
Locations (9):
- Rusk Institute, New York, New York, United States
- China (2):
  - Sichuan 81 rehabilitation center, Chengdu, Sichuan
  - China Research rehabilitation center, Beijing
- Sheba medical center, Tel Aviv, Israel
- Sunnaas rehabilitation Hospital, Nesoddtangen, Norway
- Palestinian Territories (2):
  - Betlehem arab society rehabilitation, Bethlehem, Palestine
  - El Wafa rehabilitation center, Gaza
- Petrozavodsk, Petrozavodsk, Russia
- Sahlgrenska university hospital, Gothenburgh, Sweden